CLINICAL TRIAL: NCT05209061
Title: Cellular Composition of the Human Appendix Using Single-cell RNA and Single-cell ATAC-sequencing.
Brief Title: Mapping the Human Appendix Using Single Cell Sequencing
Acronym: APPATA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bispebjerg Hospital (Other)
Collaborators: The Novo Nordisk Foundation Center for Basic Metabolic Research (Other)
Responsible Party: Principal Investigator, Jacob Antonsen, Senior Registrar, Bispebjerg Hospital
Other Study IDs: APPKOA1
Record Dates: First submitted 2022-01-12; First posted 2022-01-26 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Diabetes; Appendicitis; Inflammatory Bowel Diseases
MeSH Terms: conditions — Diabetes Mellitus; Appendicitis; Inflammatory Bowel Diseases | interventions — Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples With DNA — 1. Bloodsamples, including full blood, serum and plasma
  2. Full thickness biopsy of the appendix
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Colo-rectal cancer patients: Patients receiving right colectomy or ileo-ceacal resection for colorectal cancer
  Interventions: Other: Biopsy

INTERVENTIONS:
Other: Biopsy — Participants included in the study, will have a full thickness biopsy of the middle of the appendix taken, after the resected bowel has been removed during surgery.

SUMMARY:
The overall purpose of this study is to describe the cellular composition of the human appendix and its gene expression using scRNAseq and scATACseq methods. This will potentially provide is with a complete and detailed map of the appendix´ immunological properties and its role in neuro-endocrine/metabolic functions. Our results will be held up against current knowledge of the appendix and its role in the human body and thus hopefully expand our understanding of this organ and the consequences of its removal by appendectomy.

DETAILED DESCRIPTION:
Until recently the human appendix was viewed as a rudimentary organ without any specific function in the human body. Our current knowledge of the cellular composition of the appendix is solely based on histological examinations combined with immunohistochemical stains. These examinations have shown that the structural composition of the appendix is similar to the large intestine, with mucosa, submucosa, muscularis externa and serosa. Uniquely, the appendix has almost circumferential lymphoid follicles in the submucosa and lamina propria, and thus becomes a secondary lymphoid organ. In addition to this, the appendix contains Lieberkühn's crypts, which in contrast to the large intestine contains Paneth cells and argentaffine (enterochromaffin) neuro-endocrine cells1 2

Recently, the appendix´ role in regulation of immunologic functions has been discovered. It is believed that the great bacterial diversity in the appendix stimulates the human immune system and aids in the maturation and diversification of white blood cells, especially B-cells in the lymphoid follicles in the appendix.3 The appendix contains a larger quantity of CD5+ (B1), CD19+, Immunoglobulin-secreting IgG and secretory IgA cells compared to the large intestine. In the luminal follicle-associated epithelium, a high concentration of intra-epithelial M-cells as well as human leukocyte antigen D-related (HLA-DR) T and B cells are seen.4

The human appendix has a unique cellular composition, which plays a role in bacterial homeostasis in the large intestine5 and entero-endocrine regulation6. Furthermore, removing the appendix can drastically change incidence of certain metabolic and immune-related diseases such as type II diabetes7 and ulcerative colitis8. Despite this, only very few studies have investigated the cellular composition of the human appendix, and none of these have used single-cell (sc) RNA or DNA-sequencing to aid in our understanding of this organ.

By using scRNAseq and scATACseq (Single-cell Assay of Transposase Accessible Chromatin sequencing) we will be able to map open regions in the cell's DNA and RNA, thus providing us with a unique "map" of the cells in the appendix as well is their gene expression9-11. ScATACseq visualizes open regions in the chromatin, generating "peaks" which can then be used to map DNA motifs, such as transcription factor binding sites. With the emergence of scATACseq, chromatin accessibility is in combination with gene expression data an extremely useful resource to study cell type specific regulatory DNA interactions. To further study the immunological aspects of the appendix, we will extract immune cells from the Peyer´s plaques. Lastly, full blood will be extracted to better analyse metabolic risk factors in relation to the appendix´ metabolic cellular regulation.

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing a right or extended right-hemicolectomy for colon cancer

Patients able to read and understand danish

Patients able to give informed consent

Patients of Scandinavian ethnicity

Exclusion Criteria:

Previous large bowel resections

Suspicion pre or intraoperatively of disease in the appendix

Tumour <10cm from the appendiceal orifice.

Known inflammatory bowel disease

Immuno-modulation treatment

Neo-adjuvant chemotherapy.

< 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with verified colorectal-cancer, who have been scheduled for right colectomy or ileo-ceacal resection.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Profiling of open chromatin regions | 2 years
  Mapping of cell types, including rare cell types, using profiling of open chromatin regions. (ATAC-seq) in biopsies from the appendix
Evaluation of metabolic profile | 2 years
  Using bioimpedance, insulin and glucose measurements and CHiP-seq we will determine patient phenotype and epigenetics to evaluate their metabolic risk-profile and correlate this to cell types in the appendix

SECONDARY OUTCOMES:
Appendix biofilm | 2 years
  By sequencing bacterial DNA in our samples, we will evaluate the mucosa-associated microbiome of the appendix. This will be correlated to the two primary outcome measure

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Antonsen, MD, Principal Investigator — Bispebjerg Hospital
Locations (1):
- Bispebjerg University Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
Data in this study is based on biological samples and data from patient registry.
  These data are protected by the Danish Act on Processing of Personal Data and can be accessed through application to and approval from the Danish Data Protection Agency and the Danish Health Data Authority [https://sundhedsda tastyrelsen.dk/da/forskerservice/ansog-om-data] where the purpose and the feasibility of the intended analysis should be accounted for.

REFERENCES:
- [Background] Kooij IA, Sahami S, Meijer SL, Buskens CJ, Te Velde AA. The immunology of the vermiform appendix: a review of the literature. Clin Exp Immunol. 2016 Oct;186(1):1-9. doi: 10.1111/cei.12821. Epub 2016 Jul 19. PMID 27271818
- [Background] Somekh E, Serour F, Gorenstein A, Vohl M, Lehman D. Phenotypic pattern of B cells in the appendix: reduced intensity of CD19 expression. Immunobiology. 2000 Jan;201(3-4):461-9. doi: 10.1016/S0171-2985(00)80098-4. PMID 10776800
- [Background] Spencer J, Finn T, Isaacson PG. Gut associated lymphoid tissue: a morphological and immunocytochemical study of the human appendix. Gut. 1985 Jul;26(7):672-9. doi: 10.1136/gut.26.7.672. PMID 3874811
- [Background] Wei PL, Tsai MC, Hung SH, Lee HC, Lin HC, Lee CZ. Risk of new-onset type II diabetes after appendicectomy. Br J Surg. 2015 Sep;102(10):1267-71. doi: 10.1002/bjs.9875. Epub 2015 Jun 29. PMID 26122401
- [Background] Sahami S, Wildenberg ME, Koens L, Doherty G, Martin S, D'Haens GRAM, Cullen G, Bemelman WA, Winter D, Buskens CJ. Appendectomy for Therapy-Refractory Ulcerative Colitis Results in Pathological Improvement of Colonic Inflammation: Short-Term Results of the PASSION Study. J Crohns Colitis. 2019 Feb 1;13(2):165-171. doi: 10.1093/ecco-jcc/jjy127. PMID 30285094
- [Background] Buenrostro JD, Wu B, Chang HY, Greenleaf WJ. ATAC-seq: A Method for Assaying Chromatin Accessibility Genome-Wide. Curr Protoc Mol Biol. 2015 Jan 5;109:21.29.1-21.29.9. doi: 10.1002/0471142727.mb2129s109. PMID 25559105
- [Background] Lake BB, Codeluppi S, Yung YC, Gao D, Chun J, Kharchenko PV, Linnarsson S, Zhang K. A comparative strategy for single-nucleus and single-cell transcriptomes confirms accuracy in predicted cell-type expression from nuclear RNA. Sci Rep. 2017 Jul 20;7(1):6031. doi: 10.1038/s41598-017-04426-w. PMID 28729663
- [Background] Wagner A, Regev A, Yosef N. Revealing the vectors of cellular identity with single-cell genomics. Nat Biotechnol. 2016 Nov 8;34(11):1145-1160. doi: 10.1038/nbt.3711. PMID 27824854